CLINICAL TRIAL: NCT07395063
Title: A Single-arm, Open-label Clinical Study of Irinotecan Liposome Combined With Capecitabine, Bevacizumab and Camrelizumab as Second-line or Higher Treatment for Patients With Metastatic Colorectal Cancer
Brief Title: A Clinical Study on the Treatment of Metastatic Colorectal Cancer at the Second-line or Beyond.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-254
Record Dates: First submitted 2026-01-09; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Colorectal Cancer (CRC)
Keywords: Metastatic colorectal cancer of stage ll or higher; The treatment regimen of irinotecan liposome combined with capecitabine and camrelizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Bevacizumab; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Irinotecan liposome combined with capecitabine, bevacizumab and camrelizumab (Experimental): Zeirinotecan liposome: 60mg/m2, intravenous drip, completed within 90 minutes (±5 minutes). On the first day, administer once every 3 weeks.
  Capecitabine: 800mg/m ² orally, twice daily from day 1 to day 14, repeated every 3 weeks.
  Bevacizumab: 7.5mg/kg, intravenous infusion, day 1, once every 3 weeks; Camrelizumab: 200mg, intravenous infusion, on the first day, once every 3 weeks
  Interventions: Drug: Irinotecan liposome combined with capecitabine, bevacizumab and camrelizumab

INTERVENTIONS:
Drug: Irinotecan liposome combined with capecitabine, bevacizumab and camrelizumab — Zeirinotecan liposome: 60mg/m2, intravenous drip, completed within 90 minutes (±5 minutes). On the first day, administer once every 3 weeks.
  Capecitabine: 800mg/m ² orally, twice daily from day 1 to day 14, repeated every 3 weeks.
  Bevacizumab: 7.5mg/kg, intravenous infusion, day 1, once every 3 weeks; Camrelizumab: 200mg, intravenous infusion, on the first day, once every 3 weeks

SUMMARY:
A single-arm, open-label clinical study of irinotecan liposome combined with capecitabine, bevacizumab and camrelizumab as second-line or above treatment for patients with metastatic colorectal cancer, aiming to evaluate the efficacy and safety of irinotecan liposome combined with capecitabine, bevacizumab and camrelizumab as second-line or above treatment for patients with metastatic colorectal cancer The medication regimen is irinotecan liposome (II) + capecitabine + bevacizumab + camrelizumab until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients pathologically diagnosed with colorectal cancer;
* Received systemic treatment on the first line;
* Age: 18 to 75 years old, gender not limited.
* There must be at least one measurable lesion as the target lesion (in accordance with the RECIST v1.1 standard);
* ECOG: 0-1;
* Expected survival period ≥3 months;
* Women of childbearing age must undergo a blood pregnancy test within 3 days before randomization, and the result must be negative. They must also be willing to take appropriate contraceptive measures during the trial and for 6 months after the end of treatment. For men, it should be agreed to use appropriate methods of contraception during the study period and within 3 months after the end of treatment;
* The subjects voluntarily joined this study and signed the informed consent form.

Exclusion Criteria:

* Patients with wild-type RAS and BRAF, whose primary lesion is located in the left colorectal tract, but who have not received cetuximab as the first-line treatment
* Patients with advanced colorectal cancer who have MSI-H or dMMR
* Those with a history of other malignant diseases in the last five years, except for cured skin cancer and cervical carcinoma in situ
* For patients with a history of uncontrolled epilepsy, central nervous system diseases or mental disorders, the researcher will determine that the clinical severity may prevent them from signing the informed consent form or affect their compliance with oral medication
* Clinically severe (i.e., active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) grade II or more severe congestive heart failure, or severe arrhythmia requiring drug intervention (see Appendix 12), or a history of myocardial infarction within the last 12 months
* Those who need immunosuppressive therapy for organ transplantation
* Severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases
* The baseline blood routine and biochemical indicators of the subjects did not meet the following criteria: hemoglobin ≥90g/L; The absolute neutrophil count (ANC) is ≥1.5×109/L; Platelet count ≥100×109/L; ALT and AST≤2.5 times the normal upper limit value; ALP≤2.5 times the normal upper limit value; Serum total bilirubin <1.5 times the normal upper limit value; Serum creatinine <1 times the upper limit of normal; Serum albumin ≥30g/L
* Those known to have a deficiency of dihydropyrimidine dehydrogenase (DPD)
* Those who are allergic to any investigational drug ingredients (such as irinotecan, irinotecan liposome, capecitabine, bevacizumab and camrelizumab)
* Pregnant or breastfeeding women
* Have received any of the following treatments:

The concomitant medication contained CYP3A4, CYP2C8 strong suppressor/strong inducer or UGT1A1 strong suppressor within 2 weeks prior to randomization;Use immunosuppressants or systemic hormones for immunosuppressive purposes within 2 weeks before randomization (dose >10mg/ day, prednisone or other equivalent therapeutic hormones); <s:1> Received radiotherapy within 2 weeks prior to randomization;Undergo major surgeries (such as thoracotomy, laparotomy, etc.) within 4 weeks before randomization;The patient has received any other clinical study drug treatment within 4 weeks prior to randomization, unless it is an observational (non-interventional) clinical study or follow-up of an interventional clinical study.

- Abnormal coagulation function, with a bleeding tendency, or currently undergoing thrombolytic or anticoagulant therapy. Prophylactic use of low-dose aspirin (≤100mg/ day) and low-molecular-weight heparin (enoxaparin 40mg/ day and other low-molecular-weight heparin at equivalent doses) is permitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS） | through study completion,about 3 years
  Progression-free survival (PFS) is a measure used in clinical trials and medical research to evaluate the effectiveness of treatments, especially in oncology. It refers to the length of time during and after treatment that a patient lives with a disease without it getting worse. In other words, PFS is the duration from the start of treatment until the disease progresses or until the patient dies from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | through study completion,about 3 years
  The objective response rate (ORR) is a key endpoint used in clinical trials, particularly in oncology, to assess the effectiveness of a treatment in shrinking or eliminating tumors. It is defined as the proportion of patients in a study who achieve a partial response (PR) or a complete response (CR) to the treatment.
Duration of remission (DoR） | through study completion,about 3 years
  Duration of remission (DoR) is a critical metric in clinical oncology and hematology, particularly when evaluating the effectiveness of treatments for cancers or other diseases that can enter a state of remission. It refers to the length of time during which a patient's disease remains in remission following treatment.
Disease Control Rate (DCR） | through study completion,about 3 years
  the proportion of patients whose disease is controlled by the treatment. It includes patients who achieve a complete response (CR), partial response (PR), or stable disease (SD) after treatment.
Overall survival | through study completion,about 3 years
  OS is defined as the duration from the start of treatment or diagnosis until death from any cause. It represents the ultimate measure of a treatment's impact on patient longevity.

CONTACTS AND LOCATIONS:
Overall Officials: DEZHI LI, Principal Investigator — 4th Affiliated Hospital, School of Medicine, Zhejiang University, China

DOCUMENTS (1):
  • Study Protocol (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT07395063/Prot_000.pdf